CLINICAL TRIAL: NCT02242214
Title: REgistry of MisOprostol 200 µg Vaginal dElivery System
Acronym: REMOVE
Status: Completed | Type: Observational
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: 000188
Record Dates: First submitted 2014-09-12; First posted 2014-09-17 (Estimated); Last update posted 2015-09-16 (Estimated); Status verified 2015-09

CONDITIONS: Induction of Labour
MeSH Terms: interventions — Misoprostol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Days

GROUPS / COHORTS (1):
- Misoprostol 200 µg VDS: At the discretion of the investigator in accordance with their usual practice and consistent with the Dutch prescribing information.
  Interventions: Drug: Misoprostol

INTERVENTIONS:
Drug: Misoprostol
  Other Names: Misodel®

SUMMARY:
The design of the study is post-marketing, observational, multi-centre and open-label. The study does not provide treatment; only patients to whom misoprostol 200 µg vaginal delivery system (VDS) is prescribed may be included. All directions for medication usage and patient monitoring are solely at the discretion of the investigator in accordance with their usual practice and must be consistent with the Dutch prescribing information of misoprostol 200 µg VDS. No other (invasive) study-related interventions or measurements are done, other than the procedures routinely performed during induction of labour. No effort is expected from the study subjects. 150 patients from 20 Dutch centres will be included.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of induction of labour in women with an unfavourable cervix, from 36 weeks gestation, in whom induction is clinically indicated
* Decision made to prescribe misoprostol 200 µg VDS according to Summary of Product Characteristics (SmPC)
* Willingness and ability to provide written informed consent

Exclusion Criteria:

* Misoprostol 200 µg VDS is contraindicated according to the SmPC

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Academic and peripheral hospitals in the Netherlands
Sampling Method: Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2014-09; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Time to vaginal delivery of the neonate in hours | From insertion until vaginal delivery

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals
Locations (1):
- Isala Klinieken (there may be other sites in this country), Zwolle, Netherlands